CLINICAL TRIAL: NCT07102186
Title: Comparing the Efficacy and Safety of Adapalene Gel and Hyaluronic Acid Versus Adapalene Gel Alone in Mild to Moderate Acne Vulgaris: An Open-label Randomized Controlled Trial.
Brief Title: Efficacy and Safety of Adapalene Gel and Hyaluronic Acid Versus Adapalene Gel Alone in Mild to Moderate Acne Vulgaris
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Hebatallah Ahmed Mohamed Moustafa, Assistant professor in the clinical pharmacy and pharmacy practice department, Badr University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUC-IACUC-241117-119
Record Dates: First submitted 2025-07-21; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Acne Vulgaris
Keywords: acne vulgaris; adapalene; Hyaluronic acid; Topical Retinoids
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- adapalene gel 0.1% once daily at bedtime (Active Comparator)
  Interventions: Drug: use of adapalene gel 0.1% once daily at bedtime
- adapalene gel 0.1% once daily at bedtime and hyaluronic acid (Experimental)
  Interventions: Drug: use of adapalene gel 0.1% and hyaluronic acid at bedtime

INTERVENTIONS:
Drug: use of adapalene gel 0.1% and hyaluronic acid at bedtime — in this intervention a combination of adapalene gel 0.1% and hyaluronic acid will be used
  Arms: adapalene gel 0.1% once daily at bedtime and hyaluronic acid
Drug: use of adapalene gel 0.1% once daily at bedtime — in this intervention involves the use of adapalene gel 0.1% once daily only topically at bedtime
  Arms: adapalene gel 0.1% once daily at bedtime

SUMMARY:
Acne vulgaris affects around 85% of adolescents and young adults. Adapalene, a topical retinoid, is a common treatment but often causes irritation, leading to poor adherence. Hyaluronic acid (HA), known for its hydrating and anti-inflammatory properties, may help reduce these side effects.

This prospective, open-label, randomized controlled trial compares adapalene 0.1% gel combined with HA serum versus adapalene alone over 8 weeks in patients with mild to moderate acne. Key outcomes include acne lesion reduction, incidence and severity of side effects (erythema, dryness, scaling, stinging/burning, pruritus), and skin hydration assessed through the skin turgor test. Acne severity will be measured using the Acne Severity Index (ASI) and Investigator's Global Assessment (IGA) scale.

The study anticipates better efficacy, reduced irritation, and improved skin hydration with the combination therapy. Ethical approval was obtained, and informed consent will be secured from all participants.

DETAILED DESCRIPTION:
Acne vulgaris is a prevalent dermatological condition affecting approximately 85% of adolescents and young adults. Topical retinoids, such as adapalene, are considered a first-line treatment for mild to moderate acne due to their comedolytic, anti-inflammatory, and keratolytic properties. However, retinoid-associated irritation, including dryness, erythema, and peeling, often leads to poor adherence and treatment discontinuation.

Hyaluronic acid (HA), a naturally occurring glycosaminoglycan, is well known for its hydrating and anti-inflammatory properties. When combined with adapalene, it may improve patient adherence by reducing retinoid-induced irritation while maintaining or enhancing the therapeutic effects. While previous studies have assessed individual efficacy, there is a lack of direct comparative studies evaluating the combination of adapalene with hyaluronic acid versus adapalene alone in treating mild to moderate acne vulgaris.

The aim of this study is to compare the reduction in acne lesion count between adapalene and hyaluronic acid versus adapalene alone over 8 weeks, to evaluate differences in treatment-related adverse effects such erythema, scaling, dryness, stinging or burning, and pruritus, and to determine overall skin hydration.

This is a prospective, open-label, randomized controlled trial conducted at a dermatology clinic. Patients will be randomized into two groups: (1) adapalene 0.1% gel + hyaluronic acid serum and (2) adapalene 0.1% gel alone. The study duration will be 8 weeks with assessments at baseline and the 2nd, 4th, and 8th weeks. Patients with mild to moderate acne vulgaris who have not used topical retinoids or systemic acne treatments within the past 3 months will be included. Exclusion criteria include patients with severe acne, nodulocystic acne, secondary infections, known hypersensitivity to adapalene or hyaluronic acid, pregnant, or lactating individuals.

The acne severity index (ASI) will be assessed at baseline and at the end of the study to evaluate acne severity, considering both lesion count and distribution. The investigator's global assessment (IGA) clinical tool will be used at baseline and every 2 weeks thereafter to assess the severity of acne and monitor treatment response. It is a 5-point ordinal scale that evaluates the overall severity of acne based on lesion count, type, and inflammation. The skin turgor test will be used to assess skin hydration and the time it takes for the skin to return to its original position is observed (> 2 seconds: moderate to severe dehydration, <2 seconds, but not immediately: mild dehydration, and immediately: absent dehydration). Local tolerance to the drugs will be evaluated by using the score: 0-none; 1-mild; 2-moderate; 3-severe for erythema, scaling, dryness, stinging or burning, and pruritus at each follow-up visit.

The investigators expect a greater reduction in acne lesion counts, a lower incidence and severity of retinoid-associated irritation, and an improved skin hydration with combination therapy. Institutional Review Board (IRB) approval was obtained before initiating data collection (BUC-IACUC-241117-119). Data confidentiality will be ensured through secure storage and anonymization. Written informed consent will be obtained from all participants.

This study aims to provide clinical evidence supporting the role of hyaluronic acid in enhancing the efficacy and tolerability of adapalene in acne treatment, potentially improving patient outcomes and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate acne vulgaris who have not used topical retinoids or systemic acne treatments within the past 3 months will be included.

Exclusion Criteria:

* patients with severe acne, nodulocystic acne, secondary infections, known hypersensitivity to adapalene or hyaluronic acid, pregnant, or lactating individuals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-10-21 (Estimated); Study Completion 2025-10-21 (Estimated)

PRIMARY OUTCOMES:
Local tolerance to the drugs scale | 8 weeks
  Local tolerance to the drugs will be evaluated by using the score: 0-none; 1-mild; 2-moderate; 3-severe for erythema, scaling, dryness, stinging or burning, and pruritus at each follow-up visit. The higher the score the lower the tolerance to the drugs. Minimum score is zero and maximum score is 15.

SECONDARY OUTCOMES:
investigator's global assessment (IGA) | 8 weeks
  investigator's global assessment (IGA) clinical tool will be used at baseline and every 2 weeks thereafter to assess the severity of acne and monitor treatment response. It is a 5-point ordinal scale that evaluates the overall severity of acne based on lesion count, type, and inflammation. Only patients with score of 2 (mild) or 3 (moderate) will be enrolled and followed up
acne severity index | 8 weeks
  The acne severity index (ASI) will be assessed at baseline and at the end of the study to evaluate acne severity, considering both lesion count and distribution.The higher the score the poorer the outcomes. Minimum score is zero.
skin turgor assessment | 8 weeks
  The skin turgor test will be used to assess skin hydration and the time it takes for the skin to return to its original position is observed (> 2 seconds: moderate to severe dehydration, <2 seconds, but not immediately: mild dehydration, and immediately: absent dehydration).

CONTACTS AND LOCATIONS:
Locations (1):
- Badr university in Cairo, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol and informed consent form
Supporting Information: Study Protocol, ICF
Time Frame: 21-7-2025 till 21-10-2025
Access Criteria: data will be available via the main investigator, email: hebatallah.ahmed@buc.edu.eg